CLINICAL TRIAL: NCT03525834
Title: Phase IV, Single Arm Study of Safety and Efficacy of Everolimus in Chinese Adults With Tuberous Sclerosis Complex Who Have Renal Angiomyolipoma Not Requiring Immediate Surgery
Brief Title: Safety and Efficacy of Everolimus (Afinitor®) in Chinese Adult Patients With Angiomyolipoma Associated With Tuberous Sclerosis Complex.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001M2401
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Renal Angiomyolipoma
Keywords: TSC; tuberous sclerosis complex; AML; afinitor; everolimus; RAD001; mTOR; kidney; lymphangioleiomyomatosis; renal angiomyolipoma
MeSH Terms: conditions — Angiomyolipoma; Tuberous Sclerosis; Lymphangioleiomyomatosis | interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: Single arm, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus (Experimental): Participants targeted to receive Everolimus tablets 10 mg orally once daily for 48 weeks.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus 2.5 mg and 5 mg tablets with dosage regimen of 10 mg orally once daily.
  Other Names: RAD001, Afinitor®

SUMMARY:
The purpose of this study was to assess the safety and efficacy of everolimus (Afinitor®) in Chinese patients with renal angiomyolipoma (AML) associated with tuberous sclerosis complex (TSC).

DETAILED DESCRIPTION:
This was an open label, single arm, multi-center, Phase IV Post-Approval Commitment (PAC) study with once daily oral dose of 10 mg everolimus in participants with renal AML associated with TSC. There were three separate phases in this study: a Screening phase, an Open-label treatment phase where participants received everolimus for 48 weeks or until disease progression, and a Treatment discontinuation follow-up phase for patients who discontinue study drug for reasons other than disease progression. Every participant had an End of Treatment visit within 28 days after last dose and a safety follow-up visit 30 days after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for treatment with everolimus as per the locally approved label.
* Presence of at least one AML ≥ 3 cm in its longest diameter using CT or MRI.

Exclusion Criteria:

* AML related bleeding or embolization during the 6 months prior to enrollment.
* History of myocardial infarction, angina or stroke related to atherosclerosis.
* Impaired lung function.
* Significant hematological or hepatic abnormality.
* Any severe and/or uncontrolled medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled in 5 different sites in China.
Pre-assignment Details: Participants underwent a screening period of up to 28 days. All participants started the treatment at 10 mg orally once daily except one that started at 5 mg once daily due to a protocol deviation.
Groups:
- Everolimus: Participants targeted to receive Everolimus tablets 10 mg once daily for 48 weeks.
Period: Overall Study
Arm/Group | Everolimus
Started | 40
Completed | 39
Not Completed | 1
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian, Chinese | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Percentage of participants with AEs and SAEs including significant changes from baseline in vital signs, electrocardiograms and laboratory parameters (laboratory assessments included hematology, biochemistry, coagulation and urinalysis) qualifying and reported as AEs. The percentage of participants in each category is reported in the table.
Time Frame: From the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 52 weeks
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Participants
  AEs | 40
  Treatment-related AEs | 39
  SAEs | 6
  Treatment-related SAEs | 2

2. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) Status of Angiomyolipoma (AML) Response During Maximum Treatment Duration of 48 Weeks
Description: BOR status is the best status recorded from start of treatment until disease progression. AML response status: reduction in AML volume of at least 50% relative to screening AML. In addition, AML response have to satisfy: no new AML ≥ 1 cm in longest diameter are identified, neither kidney increases in volume by more than 20% from nadir (where nadir is the lowest kidney volume at the screening), the participant does not have any angiomyolipoma-related bleeding of grade equal or over 2 (as defined by NCI CTCAE, version 4.03).
  Up to five of the largest measurable lesions (≥ 1 cm in longest diameter) in each kidney were measured at screening via Magnetic Resonance Imaging/Computed tomography (MRI/CT) and were defined as screening AML. The sum of the volumes of these individual lesions was defined as AML volume and it was measured at each assessment during the trial. Increases in the AML volume were evidence of worsening AML, decreases were evidence of clinical response.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Participants | 28

3. Secondary Outcome: Percentage of Participants With Best Overall Response Status of Angiomyolipoma (AML) Progression During Maximum Treatment Duration of 48 Weeks
Description: AML progression status is defined as one or more of the following: an increase from nadir of 25% or more in AML volume to a value greater than screening AML (where nadir is the lowest AML volume obtained for the participant previously in the trial), the appearance of a new AML ≥ 1.0 cm in longest diameter, an increase from nadir of 20% or more in the volume of either kidney to a value greater than screening (where nadir is the lowest kidney volume obtained for the participant previously in the trial), angiomyolipoma-related bleeding grade ≥2 (as defined by NCI CTCAE, version 4.03).
  Up to five of the largest measurable lesions (≥ 1 cm in longest diameter) in each kidney were measured at screening via Magnetic Resonance Imaging/Computed tomography (MRI/CT) and were defined as screening AML. The sum of the volumes of these individual lesions was defined as AML volume and it was measured at each assessment during the trial. Increases in the AML volume were evidence of worsening AML.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Participants | 1

4. Secondary Outcome: Percentage of Participants With Severe Renal Impairment
Description: Renal impairment is defined as calculated Creatinine Clearance (CrCl) < 30 mL/min. CrCl was measured at baseline and at four other time points; only the baseline and the worst post-baseline value for every participant were counted (lowest value for CrCl).
  Creatinine clearance was estimated using the Cockcroft-Gault formula:
  creatinine clearance (mL/minute) = urine creatinine concentration (mL/dL) x volume of urine (mL/24 hour) / plasma creatinine concentration (mg/dL) x 1440 minute/24 hour
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Participants
  Baseline | 0
  Post-baseline, 48 weeks | 1

5. Secondary Outcome: Percentage of Participants With NCI CTCA Grade 3/4 Serum Creatinine
Description: NCI CTCAE grade 3/4 serum creatinine is defined as > 3.0 x upper limits of normal (ULN). Serum creatinine was measured at baseline and at four other time points; only the worst post-baseline value for every participant was counted (highest value for serum creatinine).
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 40
Participants
  Baseline | 0
  Post-baseline, 48 weeks | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 52 weeks.
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=40)
Haemorrhoids (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient psychosis (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=40)
Anaemia (Blood and lymphatic system disorders) | 8
Angular cheilitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 18
Toothache (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 6
Folliculitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 10
Blood creatinine increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 8
Blood triglycerides increased (Investigations) | 11
Creatinine renal clearance decreased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 2
Protein urine present (Investigations) | 8
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10
Epilepsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Proteinuria (Renal and urinary disorders) | 4
Menstrual disorder (Reproductive system and breast disorders) | 5
Menstruation delayed (Reproductive system and breast disorders) | 6
Menstruation irregular (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03525834/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03525834/SAP_001.pdf